CLINICAL TRIAL: NCT02429726
Title: Recombinant Adenoviral Human p53 Gene With or Without Cisplatin in Treatment of Malignant Pleural - a Phase 2, Double Blinded, Randomized, Active Controlled Study
Brief Title: Recombinant Adenoviral Human p53 Gene in Treatment of Malignant Pleural Effusion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen SiBiono GeneTech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rAd-p53-H2015002
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Malignant Pleural Effusion
Keywords: malignant pleural effusion, p53 gene therapy, cisplatin
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- rAdp53 (Experimental): 2 x 10^12 viral particles of rAdp53 gene are given in 40 ml of saline by intra-cavity infusion at day of 7, 15 and 21
  Interventions: Drug: rAdp53
- cisplatin (Active Comparator): cisplatin 40 mg in 40 ml of saline are given by intra-cavity infusion at day of 7, 15 and 21
  Interventions: Drug: Cisplatin
- rAdp53 plus cisplatin (Experimental): 2 x 10^12 viral particles of rAdp53 gene and cisplatin 40 mg in 40 ml of saline are given by intra-cavity infusion at day of 7, 15 and 21
  Interventions: Drug: rAdp53 plus cisplatin

INTERVENTIONS:
Drug: rAdp53 — Recombinant adenoviral p53 human gene will be administered by intra chest cavity infusion
  Other Names: recombinant adenoviral p53 human gene
  Arms: rAdp53
Drug: Cisplatin — Cisplatin will be administered by intra chest cavity infusion
  Arms: cisplatin
Drug: rAdp53 plus cisplatin — Recombinant adenoviral p53 human gene combined with cisplatin will be administered by intra chest cavity infusion
  Arms: rAdp53 plus cisplatin

SUMMARY:
Objective of this study is to investigate of efficacy and safety of recombinant adenoviral human p53 Gene (rAd-p53) in treatment of malignant pleural effusion, compared to cisplatin. This is a phase 2, double blinded, randomized, active controlled study.

DETAILED DESCRIPTION:
Objective of this study is to investigate of efficacy and safety of recombinant adenoviral human p53 Gene (rAd-p53) in treatment of malignant pleural effusion, compared to cisplatin. Study design: phase 2, double blinded, randomized, active controlled.Ninety patients with malignant pleural effusion, who meet the study inclusion criteria and none of exclusion criteria, will be randomized into 3 treatment groups: rAd-p53, cisplatin, and rAd-p53 combined with cisplatin. The study endpoints are objective response rate, Karnofsky score, effusion-free survival, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. histopathologically diagnosed original cancer with malignant pleural effusion;
2. 18 years or older;
3. with normal tests of hemogram, blood coagulation, liver and kidney function; 6.signed the informed consent form.
4. signed the informed consent form

Exclusion Criteria:

1. Serious blood coagulation disorder, bleeding tendency, platelet < 6 * 1000000000/L;
2. have serious heart, lung function abnormalities or severe diabetes patients;
3. active infection;
4. severe atherosclerosis;
5. AIDS patients;
6. serious thrombotic or embolic events within 6 months;
7. renal insufficiency requiring hemodialysis or peritoneal dialysis;
8. pregnant or lactating women;
9. mental disorder or disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
objective response rate | from starting study treatment to 3 months
  the rate of complete response and partial response

SECONDARY OUTCOMES:
effusion-free survival | from starting study treatment to 2 years
  effusion-free survival
Karnofsky Performance Status | from starting study treatment to 2 years
adverse events | from starting study treatment to 30 days after the last treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xi'an Jiao Tong University, Xian, Shanxi, China